CLINICAL TRIAL: NCT01003379
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, Fixed Dose Study to Assess Efficacy, Safety, and Tolerability of TC-5619 as Augmentation Therapy to Improve Cognition in Outpatients With Cognitive Dysfunction in Schizophrenia
Brief Title: TC-5619 as Augmentation Therapy to Improve Cognition in Outpatients With Cognitive Dysfunction in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-5619-238-CRD-001
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2011-12

CONDITIONS: Cognitive Dysfunction; Schizophrenia
Keywords: cognitive dysfunction; schizophrenia; Phase 2
MeSH Terms: conditions — Cognitive Dysfunction; Schizophrenia | interventions — N-(2-(pyridin-3-ylmethyl)-1-azabicyclo(2.2.2)oct-3-yl)-1-benzofuran-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC-5619 (Experimental): TC-5619 capsules will be administered once a day in a forced titration scheme at 1 mg for 4 weeks, 5 mg for 4 weeks and 25 mg for 4 weeks (12 weeks total).
  Interventions: Drug: TC-5619
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5619 — TC-5619-238 will be provided as hard gelatin capsules in strengths of 1mg, 5mg, and 25mg.
  Arms: TC-5619
Drug: Placebo — Placebo will be provided with exactly the same shape, size and appearance.
  Arms: Placebo

SUMMARY:
Schizophrenia affects approximately 1% of the population worldwide, and in about 80% of cases, it is a lifelong, disabling illness. It is a multi-dimensional disease that is associated with symptoms that have been characterized as positive, negative, and cognitive. CDS is a core feature of schizophrenia, and most individuals with schizophrenia exhibit cognitive impairment. Attention disorders, slow information processing, working memory disorders, and lack of flexibility for adaptive strategies are symptoms of cognitive impairment that have a devastating impact on the function, employment, and social status of patients with schizophrenia.

Older typical neuroleptic medications (e.g., haloperidol, fluphenazine) do not improve cognition. In fact, haloperidol has been shown to induce cognitive impairment in schizophrenic patients.

Novel atypical antipsychotics, such as risperidone, clozapine, and olanzapine, seem to produce gains in cognition. This improvement may reflect a diminution of extrapyramidal side effects of the typical high potency neuroleptics. Alternatively, it might reflect more effective symptom reduction by the novel antipsychotics, or direct cognitive enhancement through the effects of the newer agents on a variety of neurotransmitters, their receptors, and gene expression. Even when the newer antipsychotic medications improve cognition, they do not normalize it.

Presently, there are no approved therapies for CDS. However, in schizophrenic patients, nicotine improves multiple cognitive domains, including working memory and attention. Furthermore, based on a strong body of evidence ranging from genetic mapping to clinical trials, the alpha7 NNR subtype has emerged as a primary therapeutic target relevant to CDS and other core symptoms of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, per DSM-IV TR criteria, as aided by the MINI International Neuropsychiatric Interview (MINI)
* Controlled schizophrenia, on same dose of quetiapine or risperidone for no less than 2 months prior to screening
* Age 18 - 60, male or female
* Stable schizophrenia as documented by lack of psychiatric hospitalization for 2 months prior to Screening
* Clinical history of stable psychotic symptoms for 1 month prior to Screening
* Stable positive symptoms of schizophrenia for 4 weeks prior to Day 1, as shown by score ≤ 4 on PANSS for items related to delusion, hallucination, conceptual disorganization, and unusual thought content, at Screening and at Day 1
* Calgary Depression Scale for Schizophrenia score < 6
* Outpatient with stable housing, and presence of an informant who sees the subject at least 4 times weekly
* Able to understand and sign informed consent

Exclusion Criteria:

* Diagnosis of schizoaffective or schizophreniform disorders 1 year prior to Screening
* Patients at significant risk of suicide or of danger to themselves or others
* Antipsychotics other than quetiapine or risperidone, or a change in dosing of these within 2 months of Screening
* Treatment with mood stabilizers, antidepressants, or anxiolytics (short-acting hypnotics permitted)
* Treatment within 1 month using cognition-affecting agents other than the above, as listed in Appendix 3 (e.g. CNS stimulants)
* Use of other prohibited concomitant medications
* Other concomitant medications that have been changed within 1 month prior to Screening
* History within past 6 months of alcohol or illicit drug abuse
* Use of smoking cessation therapy within 1 month prior to Screening
* Tobacco users with no detectable urine cotinine level; and tobacco non-users with a detectable urine cotinine level
* Unable to comply with study procedures in opinion of investigator, including CogState battery
* History of significant other major or unstable neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, or urological disorder
* Myocardial infarction
* Seizure disorder
* Type 1 diabetes mellitus (DM); type 2 DM that requires medication (diet-controlled allowed, with HbA1C < 7.3)
* Electroconvulsive therapy within 2 months prior to Screening
* Uncontrolled hypothyroidism, vitamin B12 or folic acid deficiency
* Current TB or known systemic infection (HBV, HCV, HIV)
* Clinically significant finding on physical exam that could be a safety issue in the study
* ALT or AST levels > 2.5 times the upper limits of the laboratory reference range
* Clinically significant lab or ECG abnormality that could be a safety issue in the study, including QTcF > 450msec (males) or QtcF > 480msec (females)
* Women of child-bearing potential and men unwilling or unable to use accepted methods of birth control
* Women with a positive pregnancy test, or who are lactating
* Participation in another clinical trial in last 3 months prior to Screening
* Involvement in planning or conduct of the study by site staff

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of TC-5619 as augmentation therapy to quetiapine or risperidone, to improve cognition in stable outpatients with Cognitive Dysfunction in Schizophrenia (CDS), using the GML test of the CogState Schizophrenia Test Battery (CSTB). | Day 1 - Week 4; Week 4 - Week 8; and finally Week 8 - Week 12. There will be a 2-week follow-up period following the end of the treatment period.

SECONDARY OUTCOMES:
Assess the efficacy, safety and tolerability of TC-5619 administered adjunctively with quetiapine or risperidone, evaluate the pharmacokinetics of TC-5619 and plasma levels of quetiapine and risperidone/9-OH-risperidone. | Day 1 - Week 4; Week 4 - Week 8; and finally Week 8 - Week 12. There will be a 2-week follow-up period following the end of the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lieberman, MD, Principal Investigator — New York State Psychiatrii Institute, Columbia University
Locations (16):
- United States (7):
  - Synergy Clinical Research Center, National City, California
  - Collaborative Neuroscience Network, Inc LA County, Torrance, California
  - Altanta Center for Medical Research, Atlanta, Georgia
  - Clinical Research Institute, Wichita, Kansas
  - Neurobehavioral Reseach, Inc., Cedarhurst, New York
  - New York State Pshychiatric Institute, Columbia University, New York, New York
  - Community Clinical Research, Inc., Austin, Texas
- India (9):
  - Sravani Polyclinic and Mental Health Care Centre, Guntur, Andhra Pradesh
  - Asha Hospital, Hyderabaad, Andhra Pradesh
  - Dept. of Psychiatry, Owaisi Hospital & Research Centre, Hyderabaad, Andhra Pradesh
  - Brain Mind Behaviour Neuroscience Research Institute, Visakhapatnam, Andhra Pradesh
  - Government Hospital for Mental Care, Visakhapatnam, Andhra Pradesh
  - Adhit Khan Neuropsychiatric Centre, Mangalore, Karnataka
  - Dept. of Psychiatry, JSS University, Mysore, Karnataka
  - Mahendru Psychiatric Centre, Kanpur, Uttar Pradesh
  - Dept. of Psychiatry, CSM University, Lucknow, Uttar Pradesh